CLINICAL TRIAL: NCT02863471
Title: Open-label Pilot Phase I / II Study on Hyperthermic Intraperitoneal Chemotherapy (HIPEC) After Macroscopically Complete Resection (R0/R1) of Adenocarcinomas of the Pancreas (PanHIPEC)
Brief Title: Study on Hyperthermic Intraperitoneal Chemotherapy After Resection of Pancreascarcinoma
Acronym: PanHIPEC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PanHIPEC
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Adenocarcinomas of the Pancreas
Keywords: Pancreas; Adenocarcinoma; Hyperthermic intraperitoneal chemotherapy; HIPEC; Pancreatic surgery; Gemcitabine
MeSH Terms: conditions — Adenocarcinoma | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine (Experimental): 1000 milligram (mg)/ square meter (m²) body surface, intraperitoneal use, unique intraoperative application for 60 minutes
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Gemcitabine — 1000 milligram (mg)/square meters (m2) body surface 60 minutes (min) intraperitoneal hyperthermic lavage
  Other Names: Gemzar

SUMMARY:
In patients with peritoneal metastases of colorectal cancer could be a radical removal of all tumor foci a significantly improved survival compared to a sole systemic chemotherapy are additionally achieved by a hyperthermic intraoperative chemotherapy (HIPEC).

DETAILED DESCRIPTION:
Despite medical progress in recent years in pancreatic reach the 5-year survival rates even after radical surgical resection only 20%, which is due to high rates of local recurrence and distant metastases in the postoperative course. Due to the anatomical position of the pancreas resections are having a "wide margin" technically almost impossible, so that the tumor on postoperative preparation is often marginal forming. A further possible explanation for the high number of local recurrences, intraoperative tumor cell displacement in question.

In patients with peritoneal metastases of colorectal cancer could be a radical removal of all tumor foci a significantly improved survival compared to a sole systemic chemotherapy are additionally achieved by a hyperthermic intraoperative chemotherapy (HIPEC). Purpose of HIPEC it is to kill any remaining microscopic residual tumor or residual tumor cells free. The aim of the present phase I / II study is therefore to examine the importance of HIPEC in addition to radical resection of ductal pancreatic cancer in terms of mortality and morbidity.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Computertomographic (CT) morphologically suspected pancreatic tumor without distant metastases, with the possibility of a macroscopically complete resection residual tumor classification (R) R0 / R1 .
* Histological diagnosis of adenocarcinoma of the pancreas' in the frozen section intraoperatively
* Karnofsky Index > 70

Exclusion Criteria:

* Patients who are considered inoperable because of reduced general
* Congestive heart failure New York Heart Association (NYHA) III / IV
* Severe coronary heart disease, non-treatable arrhythmia or nonadjustable hypertension,
* Severe asthma suffering, chronic obstructive pulmonary disease (COPD)
* Renal insufficiency (serum creatinine ≥ 1.5 x of normal, or creatinine clearance <60 milliliter (ml) / minutes (min))
* Patients where the intra-operative frozen section no adenocarcinoma of the pancreas can be demonstrated
* Patients suffering from a second malignancy (within 5 years in the study of consent) except basal cell carcinoma and curative treated insitu carcinoma of the cervix
* Distant metastases (M) > 0
* Patients with a contraindication related to the present study
* Allergy or intolerance to the study drug or a substance with chemical similarity to the study medication.
* Patients under legal custodianship or incarcerated patients
* Patients that can not understand the purpose of the study due to mental, intellectual or linguistic problem
* Participation in Clinical Trials or other observation period of competing trials.
* Pregnancy, lactation
* Females of childbearing potential (FCBP) that do not agree

  * To utilize two reliable forms of contraception or practice complete abstinence from Simultaneously heterosexual contact for at least 28 days before start of treatment and for at least 28 days after administration of study treatment
  * To abstain from breastfeeding during study participation and 6 months after study treatment.
* Males that do not agree

  * to use a latex condom during any sexual contact with FCBP during participation in the study and for at least 28 days study following treatment, even if he has undergone a successful vasectomy
  * to refrain from donating semen or sperm for at least 28 days after study treatment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
30 days mortality after macroscopically complete Resection ( R0 / R1 ) of an adenocarcinoma of the pancreas in combined with hyperthermic intraperitoneal chemotherapy (HIPEC) | day 30
  Safety according to Common Terminology Criteria for Adverse Events (CTCAE) 4.0

SECONDARY OUTCOMES:
Nausea | day 30
  Safety according to Common Terminology Criteria for Adverse Events (CTCAE) 4.0
Vomiting | day 30
  Safety according to Common Terminology Criteria for Adverse Events (CTCAE) 4.0
Diarrhea | day 30
  Safety according to Common Terminology Criteria for Adverse Events (CTCAE) 4.0
Stomatitis | day 30
  Safety according to Common Terminology Criteria for Adverse Events (CTCAE) 4.0
Hair loss | day 30
  Safety according to Common Terminology Criteria for Adverse Events (CTCAE) 4.0
Neutrophilia | day 30
  Safety according to Common Terminology Criteria for Adverse Events (CTCAE) 4.0
Thrombocytopenia | day 30
  Safety according to Common Terminology Criteria for Adverse Events (CTCAE) 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Beckert, Prof. Dr., Principal Investigator — University Department of General, Visceral and TransplantSurgery Tuebingen
Locations (1):
- University Hospital, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yurttas C, Horvath P, Fischer I, Meisner C, Nadalin S, Konigsrainer I, Konigsrainer A, Beckert S, Loffler MW. A Prospective, Phase I/II, Open-Label Pilot Trial to Assess the Safety of Hyperthermic Intraperitoneal Chemotherapy After Oncological Resection of Pancreatic Adenocarcinoma. Ann Surg Oncol. 2021 Dec;28(13):9086-9095. doi: 10.1245/s10434-021-10187-8. Epub 2021 Jun 15. PMID 34131821